CLINICAL TRIAL: NCT05612373
Title: Message Offering Free Round Trip Ride-Share Ride to Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 851911-Trial C
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; behavioral science interventions; vaccination promotion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the different arms.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: As treated participants will receive text messages, there is no scope for blinding. Care providers will not be made aware of subjects' participation in the study, or assigned treatment arms. The study team will only receive data on subjects' assigned arms and outcomes at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control condition with "waiting for you" message (Experimental): This control condition will use the text message that the investigators found to be the best performing in their last mega-study of vaccine text messages to recommend a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message offering free round trip ride to the pharmacy (Experimental): This condition will use a text message offering a free round trip ride to the pharmacy to get a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages

INTERVENTIONS:
Behavioral: COVID Booster text messages — Participants will receive text messages per descriptions listed in the arms.

SUMMARY:
This experiment is part of a megastudy with a total of ten experimental conditions and a holdout control condition to which patients will be randomly assigned. The focal comparison in this experiment is between a message encouraging vaccination that provides patients with a free round trip ride-share ride to and from any pharmacy near them and a control message telling patients that an updated COVID booster vaccine is waiting for them.

ELIGIBILITY:
Exclusion Criteria:

1. The patient unsubscribed from texts before the send date and time of the patient's SMS/MMS message
2. The patient received a bivalent COVID booster before the send date and time of the patient's SMS/MMS message.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300000 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
COVID bivalent booster receipt | During the 30 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question

SECONDARY OUTCOMES:
COVID bivalent booster receipt | 60 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question
COVID bivalent booster receipt | 90 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No